CLINICAL TRIAL: NCT04398901
Title: Developmental Outcome After In Utero ZIKV Exposure in Children Without Congenital Zika Syndrome
Brief Title: Neurodevelopmental Outcomes in ZIKV-Exposed Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: Thrasher Research Fund (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sarah Mulkey, Assistant Professsor Pediatrics and Neurology, Children's National Research Institute
Other Study IDs: Pro00012759; 1R01HD102445-01 (NIH)
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Zika Virus; Congenital Zika Syndrome; Congenital Infection; Child Development
Keywords: ZIKV
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Colombia ZIKV-exposed: Seventy children in Colombia were previously enrolled as part of a fetal-neonatal neuroimaging study in 2016-2017 and were from Department of Atlantico, Colombia on the Caribbean coast. Eligible children had prior normal fetal MRI and fetal US, normal birth head circumference, normal clinical exam, no more than mild non-specific postnatal imaging findings, and are thus without findings of CZS.
  Interventions: Other: Neurodevelopmental assessments
- Colombia Non-ZIKV exposed control: The investigators will enroll 70 non-ZIKV exposed children, age 4 to 5 years, in Department of Atlántico, Colombia with birth dates prior to March 31, 2016. Based on the arrival of ZIKV to Colombia in November 2015, this date would ensure a control cohort without congenital ZIKV exposure in the first half of gestation and unlikely during any of the pregnancy.
  Interventions: Other: Neurodevelopmental assessments
- United States ZIKV-exposed: The US cohort either presented during pregnancy or after birth and sought clinical care with the Children's National Congenital Zika Program in Washington, DC and were ZIKV-exposed.
  Interventions: Other: Neurodevelopmental assessments
- United States Non-ZIKV exposed control: The investigators will enroll 32 non-ZIKV exposed children, age 4 years, in Washington, DC.
  Interventions: Other: Neurodevelopmental assessments

INTERVENTIONS:
Other: Neurodevelopmental assessments — The investigators will evaluate multiple domains of neurodevelopment at age 3, 4, 5 and 7 years using parental questionnaires and child exams. At age 7 years, the children will have a non-sedated quantitative brain MRI.

SUMMARY:
In this study the investigators will follow the neurodevelopmental outcome of children with in utero ZIKV exposure who do not have microcephaly or severe abnormalities consistent with Congenital Zika Syndrome. The ZIKV-exposed children will be compared to non-ZIKV exposed controls. Children will be assessed at age 3 and 4 years using standardized neurodevelopmental assessments. Children will also have neurodevelopmental assessment at age 5 and 7 years along with a brain MRI at age 7 years.

DETAILED DESCRIPTION:
Zika-virus (ZIKV) infection in pregnancy can result in severe brain damage in 4-12% of cases. Children exposed to ZIKV in utero during the years of 2015-2017 are now in early childhood. Children with severe neurologic injury (Congenital Zika Syndrome; CZS) have a poor developmental outcome, however the developmental outcome of apparently normal infants following in utero ZIKV-exposure is not well known. The incidence of abnormal neurodevelopmental outcome in apparently normal children with in utero ZIKV-exposure is not known.

The investigators will determine if neurodevelopmental assessment scores in children exposed to ZIKV in utero who are normal appearing differ from norms. The investigators hypothesize that ZIKV-exposed normal appearing children will have lower multi-domain developmental assessment scores compared to normative samples. The investigators hypothesize that the presence of mild postnatal non-specific cranial US findings is associated with persistent lower developmental assessment scores compared to ZIKV-exposed children who had normal cranial US and quantitative imaging will find structural and functional brain differences between ZIKV-exposed children and controls..

The investigators will perform a prospective developmental outcome study at 2 sites: 1) Department of Atlántico, Colombia through collaboration with BIOMELAB, the research center of Dr. Carlos Cure, and 2) Children's National, Washington, DC.

The objective of the study is to determine whether children who were exposed to ZIKV in utero and who do not have CZS have abnormalities in neurodevelopment during early childhood and at school age.

The primary outcome at early childhood will be neurodevelopmental assessment scores at age 3 and 4 years. Scores will be compared between Zika-exposed children and controls. The primary outcome at school age will be neurodevelopmental assessment scores at age 5 and 7 years and quantitative brain MRI at 7 years.

ELIGIBILITY:
Inclusion Criteria:

Zika-exposed cohort:

* born to mothers with Zika lab confirmation by PCR, IgM, and/or PRNT, or mother was symptomatic for Zika but infection could not be excluded due to late testing and evaluated at Children's National, Washington, DC (USA) or at BIOMELAB, Barranquilla (Colombia)
* normal fetal neuroimaging
* normal birth head circumference
* normal birth clinical exam
* no more than mild non-specific postnatal cranial ultrasound or brain MRI findings during infancy (if performed)
* able to be contacted for follow-up

Non-ZIKV exposed Controls:

* healthy
* no chronic medical conditions
* no developmental concerns
* born at term (>= 37 weeks)
* birth date prior to March 31, 2016 (Colombian controls)

Exclusion Criteria:

Zika-exposed cohort:

* another diagnosis that would impact neurodevelopment
* abnormal brain MRI (non-specific mild findings are not an exclusion criteria)

Non-ZIKV exposed controls:

* chronic medical condition with in-patient hospitalization since birth
* under care of a medical specialty provider for a chronic medical condition
* surgery with general anesthesia since birth (brief anesthesia for ear tubes, tonsillectomy, or other minor pediatric procedure is not an exclusion criteria)
* history of seizure
* abnormal vision (children wearing corrective lenses are eligible)
* abnormal hearing affecting language development
* developmental concerns expressed by caregiver
* receiving physical, occupational, speech or developmental therapy
* receiving special education services in school
* behavioral or psychological condition
* birth date March 31, 2016 or later (Colombian controls)
* preterm birth (≤36 weeks)
* planned relocation of child within 5 years and likely inability to complete study

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Zika-exposed children at 3-4 years of age (will be enrolled and studied up to age 8 years) Non-exposed controls at 4 to 5 years of age
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental assessment at age 4 years | 4 years of age
  PEDI-CAT score
Executive function | 5 and 7 years of age
  BRIEF-2 score
Motor function assessment | 5 and 7 years of age
  MABC-2 score
Brain maturation | 7 years of age
  Quantitative brain MRI volumetric measurement

SECONDARY OUTCOMES:
Motor function assessment | 4 years of age
  MABC-2 score
Intellectual ability | 5 and 7 years of age
  Age-appropriate Wechsler

CONTACTS AND LOCATIONS:
Overall Officials: Sarah B Mulkey, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (2):
- Children's National Hospital, Washington D.C., District of Columbia, United States
- Biomelab, Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time

REFERENCES:
- [Background] Mulkey SB, Peyton C, Ansusinha E, Corn E, Arroyave-Wessel M, Zhang A, Biddle C, Gutierrez C, Sorkar A, Cure A, Cure D, du Plessis AJ, DeBiasi RL, Msall ME, Cure C. Preschool neurodevelopment in Zika virus-exposed children without congenital Zika syndrome. Pediatr Res. 2023 Jul;94(1):178-184. doi: 10.1038/s41390-022-02373-5. Epub 2022 Nov 30. PMID 36446920
- [Background] Mulkey SB, Corn E, Williams ME, Peyton C, Andringa-Seed R, Arroyave-Wessel M, Vezina G, Bulas DI, Podolsky RH, Msall ME, Cure C. Neurodevelopmental Outcomes of Normocephalic Colombian Children with Antenatal Zika Virus Exposure at School Entry. Pathogens. 2024 Feb 13;13(2):170. doi: 10.3390/pathogens13020170. PMID 38392908
- [Background] Corn E, Andringa-Seed R, Williams ME, Arroyave-Wessel M, Tarud R, Vezina G, Podolsky RH, Kapse K, Limperopoulos C, Berl MM, Cure C, Mulkey SB. Feasibility and success of a non-sedated brain MRI training protocol in 7-year-old children from rural and semi-rural Colombia. Pediatr Radiol. 2024 Aug;54(9):1513-1522. doi: 10.1007/s00247-024-05964-y. Epub 2024 Jul 6. PMID 38970708
- [Background] Mulkey SB, Corn E, Williams ME, Ansusinha E, Podolsky RH, Arroyave-Wessel M, Vezina G, Peyton C, Msall ME, DeBiasi RL. Neurodevelopmental Outcomes of Preschoolers with Antenatal Zika Virus Exposure Born in the United States. Pathogens. 2024 Jun 27;13(7):542. doi: 10.3390/pathogens13070542. PMID 39057769
- [Background] Mulkey SB, Arroyave-Wessel M, Peyton C, Ansusinha E, Gutierrez C, Sorkar A, Cure A, Samper Y, Cure D, Msall ME, Cure C. Harnessing the power of telemedicine to accomplish international pediatric outcome research during the COVID-19 pandemic. J Telemed Telecare. 2024 Feb;30(2):388-392. doi: 10.1177/1357633X211063166. Epub 2021 Dec 28. PMID 34962177
- [Background] Mulkey SB, Williams ME, Peyton C, Arroyave-Wessel M, Berl MM, Cure C, Msall ME. Understanding the multidimensional neurodevelopmental outcomes in children after congenital Zika virus exposure. Pediatr Res. 2024 Aug;96(3):654-662. doi: 10.1038/s41390-024-03056-z. Epub 2024 Mar 4. PMID 38438554
- [Background] Williams ME, Corn EA, Martinez Ransanz S, Berl MM, Andringa-Seed R, Mulkey SB. Neurodevelopmental assessments used to measure preschoolers' cognitive development in Latin America: a systematic review. J Pediatr Psychol. 2024 May 16;49(5):321-339. doi: 10.1093/jpepsy/jsad089. PMID 38244996
- [Background] Mulkey SB, Andringa-Seed R, Corn E, Williams ME, Arroyave-Wessel M, Podolsky RH, Peyton C, Msall ME, Cure C, Berl MM. School-age child neurodevelopment following antenatal Zika virus exposure. Pediatr Res. 2025 Nov;98(5):1856-1863. doi: 10.1038/s41390-025-03981-7. Epub 2025 Mar 19. PMID 40108430
- [Background] Mulkey SB, DeBiasi RL. Do Not Judge a Book by Its Cover: Critical Need for Longitudinal Neurodevelopmental Assessment of In Utero Zika-Exposed Children. Am J Trop Med Hyg. 2020 May;102(5):913-914. doi: 10.4269/ajtmh.20-0197. No abstract available. PMID 32274991
- [Background] Mulkey SB, Bulas DI, Vezina G, Fourzali Y, Morales A, Arroyave-Wessel M, Swisher CB, Cristante C, Russo SM, Encinales L, Pacheco N, Kousa YA, Lanciotti RS, Cure C, DeBiasi RL, du Plessis AJ. Sequential Neuroimaging of the Fetus and Newborn With In Utero Zika Virus Exposure. JAMA Pediatr. 2019 Jan 1;173(1):52-59. doi: 10.1001/jamapediatrics.2018.4138. PMID 30476967
- [Background] Mulkey SB, Arroyave-Wessel M, Peyton C, Bulas DI, Fourzali Y, Jiang J, Russo S, McCarter R, Msall ME, du Plessis AJ, DeBiasi RL, Cure C. Neurodevelopmental Abnormalities in Children With In Utero Zika Virus Exposure Without Congenital Zika Syndrome. JAMA Pediatr. 2020 Mar 1;174(3):269-276. doi: 10.1001/jamapediatrics.2019.5204. PMID 31904798
- [Background] Mulkey SB, Ansusinha E, Cristante C, Russo SM, Biddle C, Kousa YA, Pesacreta L, Jantausch B, Hanisch B, Harik N, Hamdy RF, Hahn A, Chang T, Jaafar M, Ambrose T, Vezina G, Bulas DI, Wessel D, du Plessis AJ, DeBiasi RL. Complexities of Zika Diagnosis and Evaluation in a U.S. Congenital Zika Program. Am J Trop Med Hyg. 2021 Apr 19;104(6):2210-2219. doi: 10.4269/ajtmh.20-1256. PMID 33872214